CLINICAL TRIAL: NCT05045014
Title: Is Vestibular Dysfunction or Visuospatial Perception Affected in Individuals With Idiopathic Scoliosis
Brief Title: Evaluation of Vestibular Dysfunction or Visuospatial Perception in Individuals With Idiopathic Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate professor, Inonu University
Other Study IDs: 2021/144
Record Dates: First submitted 2021-07-14; First posted 2021-09-16 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-11

CONDITIONS: Scoliosis Idiopathic; Vestibular Function Disorder; Visuospatial/Perceptual Abilities
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Romberg test and single leg standing test will be used in balance assessment. The presence of vestibular dysfunction will be evaluated with the Utenberger test. Under the name of visual-spatial perception, spatial memory will be evaluated with the mobile application called Corsi Block Tapping, and navigation performance will be evaluated with the triangle completion task. In addition, X-ray images taken during routine follow-ups will be used to determine the location, type of curvature and Cobb angle of the scoliosis. The degree of rotation will be measured with a mobile application called Scoliodetector. Quality of life is planned to be evaluated with the Scoliosis Research Society-22 questionnaire.
  Interventions: Other: Balance assessment; Other: Unterberger test; Other: Corsi Block Tapping (mobıl app); Other: Navigation performance; Other: Cobb angle measurement; Other: Scolio Detector (mobıl app)
- Control group: Romberg test and single leg standing test will be used in balance assessment. The presence of vestibular dysfunction will be evaluated with the Utenberger test. Under the name of visual-spatial perception, spatial memory will be evaluated with the mobile application called Corsi Block Tapping, and navigation performance will be evaluated with the triangle completion task.
  Interventions: Other: Balance assessment; Other: Unterberger test; Other: Corsi Block Tapping (mobıl app); Other: Navigation performance

INTERVENTIONS:
Other: Balance assessment — Romberg test and one-leg standing test will be used.
Other: Unterberger test — During 50 steps, he will count in place with 45 degrees of hip flexion, and after 50 steps, the angle of rotation between the first position and the final position of the right foot will be measured with the help of a goniometer and the displacement distance.
Other: Corsi Block Tapping (mobıl app) — Spatial memory will be evaluated.
Other: Navigation performance — Two triangles (one equilateral, one oblique triangle, at 30°, 60° and 90° angles respectively) with route segment lengths between 150 and 300 cm will be marked on the floor and the participants will be asked to complete the task with their eyes closed. The final deviation amount will be recorded.
Other: Cobb angle measurement — It will be evaluated with the help of X-ray.
  Groups: Patient group
Other: Scolio Detector (mobıl app) — The degree of rotation will be measured with the mobile application called Scolio Detector.
  Groups: Patient group

SUMMARY:
This study was planned to investigate whether there is a visual-spatial perception disorder in individuals with idiopathic scoliosis and also to reveal its dependent/independent relationship with vestibular dysfunction.

DETAILED DESCRIPTION:
Vestibular dysfunction is thought to be associated with the etiology of patients with idiopathic scoliosis. However, there is limited data on this in the literature. However, visuospatial ability has been evaluated in the literature regarding vestibular dysfunction independent of scoliosis. In the study, it was first requested to investigate vestibular dysfunction in patients with scoliosis. However, as far as is known, there is no study in the literature on visuospatial perception investigated for vestibular dysfunction in patients with scoliosis. This study was planned to investigate whether there is a disorder related to visuospatial perception and to reveal its dependent/independent relationship with vestibular dysfunction. Based on the studies, it is planned to evaluate visuospatial (visual-spatial) perception performance in the presence/absence of vestibular dysfunction in individuals with idiopathic scoliosis. The hypothesis of the study is that vestibular function and related visual-spatial perception may be affected in individuals with idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

For the patient and control group;

* Those who do not have any other joint deformity,
* Those between the ages of 10-25,
* Individuals with good mental status Only for the experimental group
* Individuals diagnosed with idiopathic scoliosis,
* Those who have not received physiotherapy and rehabilitation for idiopathic scoliosis in the last 6 months,

Exclusion Criteria:

* Those with severe hearing and visual impairment, any neurological, orthopedic, metabolic, rheumatological disorders other than idiopathic scoliosis
* Other types of scoliosis,
* Individuals with benign paroxysmal positional vertigo, meniere, primary pathologies of the ear and a history of serious infection (ear, internal organ) will be excluded
* In healthy individuals, shoulder height difference during scanning, visual impairment, dizziness in the last 1 year, glasses wearers and individuals with a history of middle ear infection

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals with idiopathic scoliosis and healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of vestibular dysfunction-1 | 10 month
  Unterberger test will be used. Subjects will close their eyes and measure displacement in 50 steps with their shoulders flexed 90 degrees and arms extended forward.
Visual spatial perception | 10 month
  The mobile application score called Corsi Block Tapping will be recorded.
Evaluation of vestibular dysfunction-2 | 10 month
  Unterberger test will be used. Subjects will close their eyes and with their shoulders flexed 90 degrees and arms extended forward, the amount of rotation in 50 steps will be measured as an angle.

SECONDARY OUTCOMES:
Balance assessment-1 | 10 month
  Romberg test will be used. Romberg test will be recorded as (+/-) according to the individual standing with eyes closed for 30 seconds.
Navigasyon performansında | 10 month
  Two triangles (one equilateral, one oblique triangle, at 30°, 60° and 90° angles respectively) with tracktrack lengths between 150 and 300 cm will be marked on the floor and the participants will be asked to complete the task with their eyes closed. The final deviation amount will be recorded.
Quality of life assessment | 10 month
  The SRS-22r is a patient-reported outcome instrument and has a range from 1 (worst) to 5 (best). It contains 22 questions covering five domains: function, pain, self-image, mental health (each with 5 items), and satisfaction with treatment (2 items) and each item is scored from 1 to 5.
Balance assessment-2 | 10 month
  One-leg standing test will be used. The time to stand on one foot will be recorded in seconds with eyes open/closed and on hard/soft ground.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu TALU, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bigelow RT, Agrawal Y. Vestibular involvement in cognition: Visuospatial ability, attention, executive function, and memory. J Vestib Res. 2015;25(2):73-89. doi: 10.3233/VES-150544. PMID 26410672
- [Background] Le Berre M, Guyot MA, Agnani O, Bourdeauducq I, Versyp MC, Donze C, Thevenon A, Catanzariti JF. Clinical balance tests, proprioceptive system and adolescent idiopathic scoliosis. Eur Spine J. 2017 Jun;26(6):1638-1644. doi: 10.1007/s00586-016-4802-z. Epub 2016 Nov 14. PMID 27844226